CLINICAL TRIAL: NCT02999061
Title: Prevalence of Dental Caries in Preterm Birth Children Aged 2-5 Years in Primary Dentition: Across Sectional Study
Brief Title: Prevalence of Dental Caries in Preterm Birth Children Aged 2-5 Years in Primary Dentition
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ohoud Tawfig ZainElabdeen, principal investigator, Cairo University
Other Study IDs: CEBC-CU-2016-12-169
Record Dates: First submitted 2016-12-15; First posted 2016-12-21 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: PreTerm Birth
Keywords: pre-term children
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine the prevalence of dental caries in preterm birth children aged 2-5 years in primary dentition.

DETAILED DESCRIPTION:
The purpose of the study is to determine the prevalence of dental caries in preterm birth children aged 2-5 years in primary dentition.

PICO format:- Population (P) = preterm children aged 2-5 years attending Cairo University Children's Hospital "Abo El-Rish" at El-Monira, Cairo, Egypt.

Outcome (O) =prevalence of dental caries

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-5 years old.
* Presence of primary teeth only.
* Children born preterm at gestational age of 6,7 and 8 month.

Exclusion Criteria:

* Children with disability or mental disorders.
* Children with immune compromising conditions.
* Hospitalized and chronically ill children.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: population is limited to preterm birth children aged 2-5 years with primary teeth only , both genders are included.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of dental caries. | 12 month
  measured by counting the number of participants affected by dental caries/total number of study sample X100 , measurement unit is a percentage (%)

SECONDARY OUTCOMES:
Assessment of oral hygiene . | 12 month
  using a Questionnaire (binary' yes or no questions'):-
  * record child brushing habits(once or twice)
  * consumption of fluoridated water (yes/no).
  * visits to dentists (yes/no)
  * Also using a dental mirror and a probe to detect presence of plaque (plaque index) and presence of caries (dmf score).
Assessment of dietary habits | 12 month
  questionnaire (binary "yes/no questions")about the past and current feeding habits:-
  * initial feeding of the child (breast or bottle answered yes/no)
  * length of the breast feeding ( normal '0-2 years" or prolonged ">2years")
  * usage of bottle after weaning (yes/no). number of meals per day (one,two or three, answered in yes/no manner)
  * number of snacks per day (one,two or three in yes/no answers).
  * Also using a dental mirror and a probe to detect caries presence (dmf score), higher scores indicates faulty dietary habits.

CONTACTS AND LOCATIONS:
Overall Officials: Eman S Elmasry, Professor, Study Director — Cairo University; Samah M Awad, Ass.Prof., Study Director — Cairo University
Locations (1):
- Cairo University Children's Hospital "Abo El-Rish" at El-Monira, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brogardh-Roth S, Stjernqvist K, Matsson L. Dental behavioural management problems and dental caries prevalence in 3- to 6-year-old Swedish children born preterm. Int J Paediatr Dent. 2008 Sep;18(5):341-7. doi: 10.1111/j.1365-263x.2007.00884.x. PMID 18802992
- [Background] Cruvinel VR, Gravina DB, Azevedo TD, Bezerra AC, Toledo OA. Prevalence of dental caries and caries-related risk factors in premature and term children. Braz Oral Res. 2010 Jul-Sep;24(3):329-35. doi: 10.1590/s1806-83242010000300012. PMID 20877971
- [Background] Davenport ES, Litenas C, Barbayiannis P, Williams CE. The effects of diet, breast-feeding and weaning on caries risk for pre-term and low birth weight children. Int J Paediatr Dent. 2004 Jul;14(4):251-9. doi: 10.1111/j.1365-263X.2004.00557.x. PMID 15242381
- [Background] Seow WK, Lam JH, Tsang AK, Holcombe T, Bird PS. Oral Streptococcus species in pre-term and full-term children - a longitudinal study. Int J Paediatr Dent. 2009 Nov;19(6):406-11. doi: 10.1111/j.1365-263X.2009.01003.x. Epub 2009 Sep 1. PMID 19732193
- [Background] Lai PY, Seow WK, Tudehope DI, Rogers Y. Enamel hypoplasia and dental caries in very-low birthweight children: a case-controlled, longitudinal study. Pediatr Dent. 1997 Jan-Feb;19(1):42-9. PMID 9048413
- [Background] Rajshekar SA, Laxminarayan N. Comparison of primary dentition caries experience in pre-term low birth-weight and full-term normal birth-weight children aged one to six years. J Indian Soc Pedod Prev Dent. 2011 Apr-Jun;29(2):128-34. doi: 10.4103/0970-4388.84685. PMID 21911951
- [Background] Saraiva MC, Bettiol H, Barbieri MA, Silva AA. Are intrauterine growth restriction and preterm birth associated with dental caries? Community Dent Oral Epidemiol. 2007 Oct;35(5):364-76. doi: 10.1111/j.1600-0528.2006.00345.x. PMID 17822485
- [Background] Tanaka K, Miyake Y. Low birth weight, preterm birth or small-for-gestational-age are not associated with dental caries in young Japanese children. BMC Oral Health. 2014 Apr 14;14:38. doi: 10.1186/1472-6831-14-38. PMID 24731399